CLINICAL TRIAL: NCT02844361
Title: Autologous Stem-cell Transplantation Versus Conventional Chemotherapy for High Risk Waldenström Macroglobulinemia - a Prospective Multicentre Phase Ⅳ Trial From China
Brief Title: Comparison of ASCT and Conventional Chemotherapy in High Risk Waldenström Macroglobulinemia
Acronym: BDH-WM03
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015006
Record Dates: First submitted 2016-07-17; First posted 2016-07-26 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Waldenström Macroglobulinemia
Keywords: high-risk; ASCT
MeSH Terms: conditions — Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- autologous stem cell transplantation (Experimental): Patients in this group will receive BEAC(BCNU+VP-16+CTX+Ara-c) as conditioning regimen and then with autologous stem cells feedback
  Interventions: Procedure: autologous stem cell transplantation
- conventional chemotherapy (Active Comparator): Patients in this group will receive previously effective chemotherapeutic regimen as consolidation therapy
  Interventions: Drug: conventional chemotherapy

INTERVENTIONS:
Procedure: autologous stem cell transplantation — Patients in this group will receive BEAC(BCNU+VP-16+CTX+Ara-c) as conditioning regimen and then with autologous stem cells feedback
  Arms: autologous stem cell transplantation
Drug: conventional chemotherapy — Patients in this group will receive previously effective chemotherapeutic regimen as consolidation therapy
  Arms: conventional chemotherapy

SUMMARY:
The purpose of this study is to evaluate whether autologous stem cell transplantation will improve the survival of patients with high-risk Waldenström macroglobulinemia, compared with conventional chemotherapy.

DETAILED DESCRIPTION:
WM patients with partial response after introduction chemotherapy will be recommended to adopt autologous stem cell transplantation or receive conventional chemotherapy (dependent on patient's choices). After transplantation or conventional chemotherapy, maintenance therapy with rituximab or thalidomide plus prednisone will be given for less than two years.

ELIGIBILITY:
Inclusion Criteria:

1. 70 years>=Aged >=18 years
2. diagnosed with high-risk LPL/WM according to the ISSWM criteria
3. untreated or mild treated without standard regimens
4. suitable for ASCT
5. with life-expectancy more than 3 months.

Exclusion Criteria:

1. diagnosed with other malignancies outside B-NHL within one year(including active center neural system lymphoma)
2. transformed lymphoma
3. liver or renal function lesion unrelated to lymphoma
4. serious complications such as uncontrolled diabetes, gastric ulcer or other serious angiocardiopathy determined by the physician
5. HIV positive or active HBV infection or other uncontrolled systematic infection
6. clinical central nervous dysfunction
7. serious surgery within 30 days
8. pregnancy or baby nursing period or un-contracepted child-bearing period woman; 9. allergy to the trail drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
progress-free survival | up to 36 months

SECONDARY OUTCOMES:
complete remission rate | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Doc, Principal Investigator — blood disease hospital, Chinese Academic Medical School
Locations (1):
- Shuhua Yi, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided
dependent on the local law